CLINICAL TRIAL: NCT01318967
Title: MRI for the Non-invasive Determination of Renal Blood Flow and Renal Oxygenation
Brief Title: Measurement of Kidney Blood Flow and Oxygen Levels by MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00010832
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Chronic Kidney Disease
Keywords: Renal blood flow; Regional renal blood flow; MRI
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PAH (Placebo Comparator): PAH measure of renal blood flow is first performed on subjects prior to administration of furosemide
  Interventions: Other: Placebo
- MRI after furosemide (Active Comparator): After the PAH measurement is complete, subjects receive 20 mg furosemide and undergo BOLD MRI to estimate renal blood flow
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Renal blood flow is measured after the administration of 20 mg of furosemide during MRI scan only.
  Other Names: Lasix
  Arms: MRI after furosemide
Other: Placebo
  Arms: PAH

SUMMARY:
Comparison of renal blood flow measurements by PAH clearance and MRI

DETAILED DESCRIPTION:
The traditional measurement of renal blood flow in ml/min involves the collection of multiple blood and urine samples after an infusion of a drug called para-aminohippurate (PAH) is given. In this study, the investigators determine the ability of MRI to estimate renal blood flow. The primary hypothesis is that renal blood flow as measured by PAH clearance is similar to renal blood flow as estimated by MRI. The measurements by PAH clearance and MRI are both performed on the same day.

ELIGIBILITY:
Inclusion Criteria:

In this study, the investigators will enroll 16 men and women aged ≥ 18 years with Stage II - V chronic kidney disease (CKD). In addition, the investigators will enroll 4 subjects with a glomerular filtration rate (GFR) of greater than 60 ml/min who do not have any evidence of CKD.

Exclusion Criteria:

This study excludes those not suitable for MRI or for the interventional pharmacologic procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rocco, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Furosemide: With and without furosemide
  Furosemide: Renal blood flow is measured before and after the administration of 20 mg of furosemide.
Period: Overall Study
Arm/Group | Furosemide
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Furosemide
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Renal Blood Flow of the Kidney by the PAH Method
Description: Renal blood flow is estimated by the PAH method.
Time Frame: Renal blood flow is estimated over 1 hour by PAH
Measure: Mean (Full Range); unit: ml/min
Groups:
- Furosemide: With and without furosemide
  Furosemide: Renal blood flow is measured before and after the administration of 20 mg of furosemide.
  Renal blood flow is measured by PAH method and by MRI method
Arm/Group | Furosemide
Number analyzed (Participants) | 10
ml/min | 190 [47 to 342]

2. Secondary Outcome: Measurement of Regional Blood Oxygenation by MRI
Description: Estimate of renal blood flow by using MRI scans before and after the administration of furosemide
Time Frame: One measure after furosemide (day 1)
Measure: Mean (Full Range); unit: ml/min
Arm/Group | MRI After Furosemide
Number analyzed (Participants) | 10
ml/min | 300 [69 to 620]

ADVERSE EVENTS:
Arm/Group | Furosemide
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No